CLINICAL TRIAL: NCT01146951
Title: A Placebo-Controlled, Double-Blind Comparative Study of E2080 in Lennox-Gastaut Syndrome Patients
Brief Title: A Placebo-Controlled, Double-Blind Comparative Study of E2080 in Lennox-Gastaut Syndrome Patients (Study E2080-J081-304)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2080-J081-304
Record Dates: First submitted 2010-06-14; First posted 2010-06-22 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Epilepsy; Seizures
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Seizures | interventions — rufinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rufinamide (E2080) (Experimental)
  Interventions: Drug: Rufinamide (E2080)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rufinamide (E2080) — Rufinamide tablets administered orally twice daily after breakfast and dinner. Treatment was divided into a Dose Titration Period (2 weeks) and a Dose Maintenance Period (10 weeks). As a general rule, the dose was increased by 1 step every 2 days until it reached the target maintenance dose determined by body weight at the start of the Observation Period.
  Target maintenance dose:
  15.0 - 30.0 kg: 1000 mg/day (5 tablets each in the morning and evening) 30.1 - 50.0 kg: 1800 mg/day (4 tablets in the morning and 5 in the evening) 50.1 - 70.0 kg: 2400 mg/day (6 tablets each in the morning and evening) >= 70.1 kg: 3200 mg/day (8 tablets each in the morning and evening)
  Other Names: E2080
  Arms: Rufinamide (E2080)
Drug: Placebo — Rufinamide Matching Placebo tablets administered orally twice daily after breakfast and dinner for a total of 12 weeks.
  Arms: Placebo

SUMMARY:
To confirm that the combination therapy of rufinamide has superior efficacy compared to placebo in patients with Lennox-Gastaut syndrome.

ELIGIBILITY:
Inclusion criteria

1. Participants who are diagnosed as Lennox-Gastaut syndrome with tonic/atonic seizures and atypical absence seizures (A history of atypical absence seizures will also be incorporated).
2. Participants who had a slow spike-and-wave pattern in an electroencephalogram within 6 months prior to the enrollment for the Observation Period.
3. Participants who had at least a total of 90 seizures in the 28 days prior to the enrollment for the Observation Period.
4. Participants who have been on 1 - 3 anti-epileptic drugs from 28 days prior to the enrollment for the Observation Period and have not changed the type of the anti-epileptic drugs.
5. Participants who have not changed the type nor the dose or administration of the anti-epileptic drugs they are taking in the Observation Period.

Exclusion criteria;

1. Participants who had a history of generalized tonic-clonic status epilepticus within baseline.
2. Participants who received drug therapy at least 4 times to be rescued from status epilepticus within baseline.
3. Participants who had a history of hypoxia which needed emergency resuscitation within 12 months prior to the Treatment Period.
4. Participants who were on a ketogenic diet or have received adrenocorticotropic hormone (ACTH) therapy or Vitamin B6 therapy within 6 months prior to the Treatment Period.
5. Participants who had a history of suicide attempt within the 1 year prior to the Treatment Period.
6. Participants who had a history of or has an allergy to triazole compound.
7. Participants who have clinically significant electrocardiogram abnormalities at baseline.
8. Participants who are pregnant, who may be pregnant, who are lactating or who wish to be pregnant.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Takano, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (23):
- Japan (23):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Yokohama, Kanagawa
  - Goshi-shi, Kumamoto
  - Iwamuma-shi, Miyagi
  - Omura-shi, Nagasaki
  - Nara, Nara
  - Niigata, Niigata
  - Yufu-shi, Oita Prefecture
  - Okayama, Okayama-ken
  - Neyagawa, Osaka
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Moriya-shi, Shiga
  - Shizuoka, Shizuoka
  - Kodaira-shi, Tokyo
  - Kokubunji-shi, Tokyo
  - Shinjuku-ku, Tokyo
  - Toyoma-shi, Toyama

REFERENCES:
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- [Derived] Panebianco M, Prabhakar H, Marson AG. Rufinamide add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Nov 8;11(11):CD011772. doi: 10.1002/14651858.CD011772.pub3. PMID 33179247

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of n= 66 who started Observation Period, 7 discontinued from study. Primary reasons were deviation of the inclusion/ exclusion criteria (n=5), untoward event before study treatment (n=1) & other (n=1). Of 59 participants, 58 were included in full analysis set (FAS). 1 participant (E2080 group) was excluded due to inappropriate diagnosis of disease.
Groups:
- Rufinamide (E2080): Rufinamide : Rufinamide tablets administered orally twice daily after breakfast and dinner. Treatment was divided into a Dose Titration Period (2 weeks) and a Dose Maintenance Period (10 weeks). As a general rule, the dose was increased by 1 step every 2 days until it reached the target maintenance dose determined by body weight at the start of the Observation Period.
  Target maintenance dose:
  15.0 - 30.0 kg: 1000 mg/day (5 tablets each in the morning and evening) 30.1 - 50.0 kg: 1800 mg/day (4 tablets in the morning and 5 in the evening) 50.1 - 70.0 kg: 2400 mg/day (6 tablets each in the morning and evening) >= 70.1 kg: 3200 mg/day (8 tablets each in the morning and evening)
- Placebo: Placebo : Rufinamide Matching Placebo tablets administered orally twice daily after breakfast and dinner for a total of 12 weeks.
Period: Overall Study
Arm/Group | Rufinamide (E2080) | Placebo
Started | 29 | 30
Completed | 25 | 29
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Population: One subject from the Rufinamide (E2080) group was excluded from the FAS because of the inappropriate diagnosis of the disease, dropping the total number from 29 to 28 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rufinamide (E2080) | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (7.1) | 13.9 (6.1) | 14.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Tonic-Atonic Seizure Frequency From Baseline (Per 28 Days)
Description: The sum of the frequencies of tonic seizures and atonic seizures was defined as the "tonic-atonic seizure frequency" and the percent change in tonic-atonic seizure frequency per 28 days was assessed. The percent change in tonic-atonic seizure frequency was calculated using the tonic-atonic seizure frequency per 28 days of the Observation Period as the baseline and the tonic-atonic seizure frequency per 28 days of the Treatment Period as the post-treatment value. Percentage change in tonic - atonic seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline].
  The frequency of epileptic seizures was recorded in the seizure diary by the recorder. Seizure frequency was counted based on the classification established by the International League Against Epilepsy (ILAE). The diary recorder monitored the participant and recorded the seizure diary in a consistent manner, and continued these practices throughout the study period.
Time Frame: Baseline (28 day observational period) and End of Treatment (28 day treatment period)
Population: Full analysis set (FAS) is defined as participants who were registered for the Treatment Period and excludes those listed below.
  Participants who did not meet the inclusion criterion related the target disease, participants who did not take the study drug, participants without any evaluable efficacy data after the start of study treatment.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Rufinamide (E2080) | Placebo
Number analyzed (Participants) | 28 | 30
Percent Change | -24.20 [-93.5 to 27.2] | -3.25 [-81.6 to 151.9]
Statistical Analysis 1: Comparison: Rufinamide (E2080) vs Placebo; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -26.65, 90% CI 2-sided [-40.30 to -11.80]

2. Secondary Outcome: Number of Participants Achieving a 50% Reduction in Tonic-atonic Seizure Frequency
Description: 50% Responder Rate in Tonic-Atonic Seizure Frequency was presented as the number of participants who achieved a 50% reduction in tonic-atonic seizure frequency.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rufinamide (E2080) | Placebo
Number analyzed (Participants) | 28 | 30
Participants
  Yes (50% Reduction Achieved) | 7 | 2
  No | 21 | 28
Statistical Analysis 1: Comparison: Rufinamide (E2080) vs Placebo; Test type: Superiority or Other; p = 0.074, Fisher's exact test

3. Secondary Outcome: Percent Change in Total Seizure Frequency (Per 28 Days)
Description: Percent change in the total seizure frequency (per 28 days) was calculated using the total seizure frequency per 28 days of the Observation Period as the baseline and the total seizure frequency per 28 days of the Treatment Period as the post-treatment value. Percentage change in total seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline].
Time Frame: Baseline (28 day observational period) and End of Treatment (28 day treatment period)
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Rufinamide (E2080) | Placebo
Number analyzed (Participants) | 28 | 30
Percent Change | -32.90 [-87.3 to 15.4] | -3.05 [-52.2 to 133.0]
Statistical Analysis 1: Comparison: Rufinamide (E2080) vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -33.30, 90% CI 2-sided [-47.10 to -17.00]

4. Secondary Outcome: Percentage Change in the Frequency of Seizures Other Than Tonic-atonic Seizures (Per 28 Days)
Description: Percent change in the frequency of seizures other than tonic-atonic seizures (per 28 days) was calculated using the total seizure frequency per 28 days of the Observation Period as the baseline and the total seizure frequency per 28 days of the Treatment Period as the post-treatment value. Percentage change in total seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline].
  Seizures analyzed other than tonic-atonic seizures included:
  Partial seizure freq. (frequency), Absence seizure, Atyp. (atypical) absence seizure, Myoclonic seizure, Clonic seizure, Tonic seizure, Tonic-clonic seizure, Atonic seizure, & Uncla. (unclassified) epileptic seizure.
  The frequency of epileptic seizures was recorded in the diary by the recorder. Seizure frequency was counted based on the classification established by the International League Against Epilepsy (ILAE). The diary recorder monitored the participant and recorded the seizure diary in a consistent manner.
Time Frame: Baseline (28 day observational period) and End of Treatment (28 day treatment period)
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Rufinamide (E2080) | Placebo
Number analyzed (Participants) | 28 | 30
Percent change
  Partial Seizure Freq. % Change (n=4,6) | -52.20 [-96.2 to -26.3] | 4.5 [-28.2 to 35.9]
  Absence Seizure Freq. % Change (n=1,0) | 3.40 [3.4 to 3.4] | NA [NA to NA] — n=0 participants with absence seizures analyzed in Placebo arm
  Atyp. Absence Seizure Freq. % Change (n=12,19) | -59.00 [-100.0 to 107.1] | -21.10 [-83.2 to 253.5]
  Myoclonic Seizure Freq. % Change (n=10,10) | -52.35 [-100.0 to 53.3] | 6.60 [-46.1 to 270.0]
  Clonic Seizure Freq. % Change (n=1,0) | -81.20 [-81.2 to -81.2] | NA [NA to NA] — n=0 participants with clonic seizures analyzed in Placebo arm
  Tonic Seizure Freq. % Change (n=28,28) | -24.20 [-92.6 to 42.8] | -3.60 [-83.8 to 274.8]
  Tonic-clonic Seizure Freq. % Change (n=2,10) | -57.35 [-100.0 to -14.7] | 2.35 [-75.8 to 450.0]
  Atonic Seizure Freq. % Change (n=10,12) | -63.10 [-100.0 to 68.8] | -6.10 [-100.0 to 2195.7]
  Uncla. Epileptic Seizure Freq. % Change (n=1,0) | -88.70 [-88.7 to -88.7] | NA [NA to NA] — n=0 participants with unclassified epileptic seizures analyzed in Placebo arm
Statistical Analysis 1: Comparison: Rufinamide (E2080) vs Placebo; Analysis for Partial Seizure Frequency; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -57.15, 90% CI 2-sided [-104.50 to -17.30]
Statistical Analysis 2: Comparison: Rufinamide (E2080) vs Placebo; Analysis of atypical absence seizure frequency; Test type: Superiority or Other; p = 0.128, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -28.65, 90% CI 2-sided [-72.00 to 0.90]
Statistical Analysis 3: Comparison: Rufinamide (E2080) vs Placebo; Analysis for myoclonic seizure frequency; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -54.35, 90% CI 2-sided [-126.60 to -15.40]
Statistical Analysis 4: Comparison: Rufinamide (E2080) vs Placebo; Analysis of tonic seizure frequency; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -23.20, 90% CI 2-sided [-40.70 to -5.60]
Statistical Analysis 5: Comparison: Rufinamide (E2080) vs Placebo; Analysis for Tonic-clonic seizure frequency; Test type: Superiority or Other; p = 0.107, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -71.40, 90% CI 2-sided [-464.70 to 30.50]
Statistical Analysis 6: Comparison: Rufinamide (E2080) vs Placebo; Analysis of Atonic seizure frequency; Test type: Superiority or Other; p = 0.221, Wilcoxon (Mann-Whitney); Hodges-Lehmann method = -52.10, 90% CI 2-sided [-89.10 to 10.80]

5. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: CGIC in participants with Lennox-Gastaut Syndrome (LGS) relative to placebo was presented as number of participants in each category at the final assessment (last observation carried forward [LOCF]) & at Week 12 of the Treatment Period. The investigator assessed the CGIC by comparing the participants' condition during the 4 weeks immediately before the completion (or discontinuation [d/c]) of the Treatment Period to his/her condition during the 4-week Observation Period (for participants who d/c'd the study during the Treatment Period, the CGIC was assessed by comparing the participant's condition from the start to discontinuation of the study treatment to his/her condition during the 4-week Observation Period).
  The CGIC was assessed according to the following 7-grade scale based on the frequency & severity of seizures, AEs, and overall conditions of daily life.
  Markedly improved, Improved, Slightly improved, Unchanged, Slightly worsened, Worsened, Markedly worsened.
Time Frame: Up to Week 12 of the treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rufinamide (E2080) | Placebo
Number analyzed (Participants) | 28 | 30
participants
  Week 12: Markedly improved (n=25, 29) | 0 | 0
  Week 12: Improved (n=25, 29) | 9 | 0
  Week 12: Slightly Improved (n=25, 29) | 4 | 9
  Week 12: Unchanged (n=25, 29) | 10 | 18
  Week 12: Slightly Worsened (n=25, 29) | 1 | 1
  Week 12: Worsened (n=25, 29) | 1 | 1
  Week 12: Markedly Worsened (n=25, 29) | 0 | 0
  LOCF: Markedly Improved (n=28, 30) | 3 | 0
  LOCF: Improved (n=28, 30) | 9 | 0
  LOCF: Slightly Improved (n=28, 30) | 4 | 9
  LOCF: Unchanged (n=28, 30) | 10 | 19
  LOCF: Slightly Worsened (n=28, 30) | 1 | 1
  LOCF: Worsened (n=28, 30) | 1 | 1
  LOCF: Markedly Worsened (n=28, 30) | 0 | 0
Statistical Analysis 1: Comparison: Rufinamide (E2080) vs Placebo; Analysis of Week 12 of the Treatment Period; Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rufinamide (E2080) vs Placebo; Analysis of final assessment (LOCF); Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From date of first dose until date of last dose of study treatment, up to approximately 1 year 2 months
Description: Treatment-emergent adverse events and treatment-emergent serious adverse events were reported for the safety analysis set, which consisted of participants who registered for the Treatment Period and excludes participants who did not take study drug and those without any evaluable safety data after the start of study treatment.
Arm/Group | Rufinamide (E2080) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/30
Other Adverse Events (participants affected / at risk) | 27/29 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (E2080) (N=29) | Placebo (N=30)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (E2080) (N=29) | Placebo (N=30)
Hypothyroidism (Endocrine disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Dental Caries (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4
Bronchitis (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Blood Pressure Decreased (Investigations) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 8 | 5
Somnolence (Nervous system disorders) | 6 | 2
Autism (Nervous system disorders) | 1 | 0
Complex Partial Seizures (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0
Tonic Convulsion (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Stereotypy (Psychiatric disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Heat Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other